CLINICAL TRIAL: NCT01876212
Title: A Randomized Phase 2 Pilot Study of Type I-Polarized Autologous Dendritic Cell Vaccines Incorporating Tumor Blood Vessel Antigen (TBVA)-Derived Peptides in Combination With Dasatinib in Patients With Metastatic Melanoma
Brief Title: Dendritic Cell Vaccines + Dasatinib for Metastatic Melanoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Walter J. Storkus (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor-Investigator, Walter J. Storkus, Associate Professor of Medicine, Clinical & Translational Science, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 12-048; R01CA169118 (NIH); UPCI 12-048 (Other: University of Pittsburgh Cancer Institute)
Record Dates: First submitted 2013-06-10; First posted 2013-06-12 (Estimated); Results first posted 2019-08-06 (Actual); Last update posted 2019-08-22 (Actual); Status verified 2019-08

CONDITIONS: Metastatic Melanoma
Keywords: melanoma; metastatic; vaccine; BRAF
MeSH Terms: conditions — Melanoma; Neoplasm Metastasis | interventions — lentiviral minigene vaccine of COVID-19 coronavirus; Dasatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Vaccine + dasatinib (Experimental): Patients will start vaccine on cycle 1, day 1 and dasatinib on cycle 2, day 1 (week 5).
  All patients will receive dasatinib at a starting dose of 70 mg twice daily by mouth in the outpatient setting. Dasatinib will be supplied as 50 mg and 20 mg tablets. Patients will take 1 of the 50 mg tablets and 1 of the 20 mg tablets twice daily, approximately every 12 hours, at the same time each day.
  The DC vaccine will be administered by a single intradermal injection of approximately 10e7 cells, with all the DCs being administered on days 1 and 15 of each cycle. The intradermal administration will be in the vicinity of the four nodal drainage groups of the four extremities.
  Interventions: Biological: DC vaccine; Drug: Dasatinib
- Vaccine + dasatinib from cycle 1 (Experimental): Patients will start vaccine on cycle 1, day 1 and dasatinib on cycle 1, day 1.
  All patients will receive dasatinib at a starting dose of 70 mg twice daily by mouth in the outpatient setting. Dasatinib will be supplied as 50 mg and 20 mg tablets. Patients will take 1 of the 50 mg tablets and 1 of the 20 mg tablets twice daily, approximately every 12 hours, at the same time each day.
  The DC vaccine will be administered by a single intradermal injection of approximately 10e7 cells, with all the DCs being administered on days 1 and 15 of each cycle. The intradermal administration will be in the vicinity of the four nodal drainage groups of the four extremities.
  Interventions: Biological: DC vaccine; Drug: Dasatinib

INTERVENTIONS:
Biological: DC vaccine
  Other Names: Type 1-polarized, autologous, DC vaccines incorporating tumor blood vessel antigen (TBVA)-derived peptides
Drug: Dasatinib
  Other Names: BMS-354825; Sprycel

SUMMARY:
Current therapeutic approaches available for patients with advanced-stage melanoma remain inadequate, and existing approaches including those involving immunotherapy with cytokines and/or targeted strategies have resulted in disappointingly low rates of durable and complete responses. Correcting immune dysfunction in advanced-stage melanoma patients using tyrosine-kinase inhibitor (TKI) such as dasatinib is proposed to relicense the patient's immune system to respond optimally to specific immunization. The integration of antigens expressed by tumor-associated blood vessel cells provides a means to selectively target the genetically-/antigenically-heterogeneous population of tumor cells in the advanced-stage melanoma patient.

This is a single-center, prospective randomized Phase 2 trial evaluating the activity, safety and immune effects of dasatinib given in combination with an autologous type-1 polarized Dendritic Cell (αDC1) vaccine. The current trial represents a randomized Phase 2 study to determine the activity and safety of intradermal (id) administration of αDC1s loaded with a mixture of six TBVA-derived peptides at the time of, or immediately after, an initial therapy cycle with the TKI dasatinib.

Dasatinib will be administered at the standard dose and schedule recommended by the FDA (70 mg BID). The autologous type-I DC vaccine will be administered either prior to, or concomitant with, the initiation of dasatinib administration. All patients will receive dasatinib at a starting dose of 70 mg twice daily by mouth in the outpatient setting approximately every 12 hours, at the same time each day.

The DC vaccine will be administered by a single intradermal injection of approximately 10e7 cells, with all the DCs being administered on days 1 and 15 of every cycle on an outpatient basis in the University of Pittsburgh Clinical and Translational Research Center (UPCI-CTRC).

Patients on Arm A will start dasatinib administration on cycle 2, day 1 (week 5), while those patients in Arm B will start dasatinib administration on cycle 1, day 1 (week 1).

Men and women at least 18 years of age must be HLA-A2+ and have histologically confirmed melanoma that is metastatic (Stage IV) or unresectable Stage IIIB/C and for which standard curative or palliative measures do not exist or are no longer effective.

Note: The outcome measures and time frames (previously) described in the PRS protocol record have been revised and articulated in the results section, to more accurately describe and represent the stated per-protocol investigations and endpoints, quantitatively.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be HLA-A2+ and have histologically confirmed melanoma that is metastatic (Stage IV) or unresectable Stage IIIB/C and for which standard curative or palliative measures do not exist or are no longer effective.
* Patients must have measurable disease by RECIST 1.1, defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded for non-nodal lesions and short axis for nodal lesions) as ≥ 20 mm with conventional techniques or as ≥ 10 mm with spiral CT scan, MRI, or calipers by clinical exam. See Section 11 for the evaluation of measurable disease.
* Patients should have at least 2 subcutaneous, intracutaneous, and accessible tumor deposits, lymph node or other site available for biopsy purposes. Patients that have one biopsiable site that can be amenable to 2 biopsies (pre- and post-) will be considered eligible.
* Prior chemotherapy, immunotherapy, or targeted therapy is allowed as long as it did not include dasatinib.
* Age ≥ 18 years. Because no dosing or adverse event data are currently available on the use of dasatinib in patients < 18 years of age, children are excluded from this study, but will be eligible for future pediatric trials.
* ECOG performance status ≤ 2 (Karnofsky ≥ 60%, see Appendix A).
* Life expectancy of greater than 12 weeks.
* Patients must have normal organ and marrow function as defined below:

  * Leukocytes ≥ 3,000/µL
  * absolute neutrophil count ≥ 1,500/µL
  * absolute lymphocyte count ≥ 500/µL
  * platelets ≥ 100,000/µL
  * total bilirubin within normal institutional limits
  * AST(SGOT)/ALT(SGPT) ≤ 2.5 X institutional upper limit of normal
  * Creatinine ≤ 2.0 X institutional upper limit of normal
* Serum magnesium, potassium and adjusted (or ionized) calcium ≥ the institutional lower limit of normal. (Supplementation of electrolytes prior to screening is allowed).
* Sexually active women and men of childbearing potential must agree to use an effective method of birth control during the course of the study and for up to 3 months following the last dose of the study drug, in a manner such that risk of pregnancy is minimized. Surgical sterilization, intrauterine device or barrier method (e.g. condom and/or diaphragm with spermicidal agents) are acceptable forms of birth control. Women of childbearing potential must have a negative pregnancy test (serum) within 7 days prior to treatment. A pregnancy test is not required for registration. Women who have not menstruated for more than 2 years will be considered postmenopausal, thus not of childbearing potential.
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Patients who have had chemotherapy or radiotherapy within 4 weeks (6 weeks for nitrosoureas or mitomycin C) prior to entering the study or those who have not recovered from adverse events due to agents administered more than 4 weeks earlier.
* Patients with documented c-KIT mutations.
* Patients who are receiving any other investigational agents.
* Patients with known active brain metastases should be excluded. Patients with treated brain metastases with documented stability for 4 weeks are eligible.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to dasatinib or any of the components of the vaccine being administered as part of this study.
* Women who are pregnant or nursing/breastfeeding.
* History of significant bleeding disorder unrelated to cancer, including:

  * Diagnosed congenital bleeding disorders (e.g., von Willebrand's disease)
  * Diagnosed acquired bleeding disorder within one year (e.g., acquired anti-factor VIII antibodies)
* Patients currently taking medications that inhibit platelet function (i.e., aspirin, dipyridamole, epoprostenol, eptifibatide, clopidogrel, cilostazol, abciximab, ticlopidine, and any non-steroidal anti-inflammatory drug) because of a potential increased risk of bleeding from dasatinib.
* Patients currently taking anticoagulants (warfarin, heparin/low molecular weight heparin [e.g., danaparoid, dalteparin, tinzaparin, enoxaparin]) because of a potential increased risk of bleeding from dasatinib.
* Diagnosis of unstable angina or myocardial infarction within 6 months of study entry.
* Patients currently taking one or more of the following drugs that are generally accepted to have a risk of causing Torsades de Pointes:

  * quinidine, procainamide, disopyramide
  * amiodarone, sotalol, ibutilide, dofetilide
  * erythromycins, clarithromycin
  * chlorpromazine, haloperidol, mesoridazine, thioridazine, pimozide
  * cisapride, bepridil, droperidol, methadone, arsenic, chloroquine, domperidone, halofantrine, levomethadyl, pentamidine, sparfloxacin, lidoflazine.
* Diagnosed or suspected congenital long QT syndrome.
* Prolonged QTc interval on pre-entry electrocardiogram (> 450 msec) within 30 days prior to study registration.
* Any history of clinically significant ventricular arrhythmias (such as ventricular tachycardia, ventricular fibrillation, or Torsades de pointes)
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* HIV-positive patients on combination antiretroviral therapy are ineligible because of the potential for pharmacokinetic interactions with dasatinib. In addition, these patients are at increased risk of lethal infections when treated with marrow-suppressive therapy. Appropriate studies will be undertaken in patients receiving combination antiretroviral therapy when indicated.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2014-05-16 (Actual); Primary Completion 2018-07-11 (Actual); Study Completion 2019-07-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Kirkwood, MD, Principal Investigator — University of Pittsburgh Cancer Institute (UPCI)
Locations (1):
- Hillman Cancer Center, Pittsburgh, Pennsylvania, United States

REFERENCES:
- [Derived] Storkus WJ, Maurer D, Lin Y, Ding F, Bose A, Lowe D, Rose A, DeMark M, Karapetyan L, Taylor JL, Chelvanambi M, Fecek RJ, Filderman JN, Looney TJ, Miller L, Linch E, Lowman GM, Kalinski P, Butterfield LH, Tarhini A, Tawbi H, Kirkwood JM. Dendritic cell vaccines targeting tumor blood vessel antigens in combination with dasatinib induce therapeutic immune responses in patients with checkpoint-refractory advanced melanoma. J Immunother Cancer. 2021 Nov;9(11):e003675. doi: 10.1136/jitc-2021-003675. PMID 34782430

RESULTS

PARTICIPANT FLOW:
Groups:
- Vaccine (Cycle 1, Day 1) + Dasatinib (Cycle 2, D1): Patients received vaccine on treatment Cycle 1, Day 1, and dasatinib beginning on treatment Cycle 2, Day 1 (week 5).
  All patients received dasatinib at a starting oral dose of 70 mg twice daily, and dasatinib as (1) 50 mg and (1) 20 mg tablets twice daily (each 12 hours).
  The DC vaccine was administered by a single intradermal injection of approximately 10^7 cells (in the vicinity of the four nodal drainage groups of the four extremities) , on days 1 and 15 of each cycle.
- Vaccine + Dasatinib (Cycle 1, D1): Patients received both vaccine and dasatinib beginning on treatment Cycle 1, Day 1.
  All patients received dasatinib at a starting oral dose of 70 mg twice daily, and dasatinib as (1) 50 mg and (1) 20 mg tablets twice daily (each 12 hours).
  The DC vaccine was administered by a single intradermal injection of approximately 10^7 cells (in the vicinity of the four nodal drainage groups of the four extremities) , on days 1 and 15 of each cycle.
Period: Overall Study
Arm/Group | Vaccine (Cycle 1, Day 1) + Dasatinib (Cycle 2, D1) | Vaccine + Dasatinib (Cycle 1, D1)
Started | 9 | 6
Completed | 9 | 6
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Vaccine (Cycle 1, Day 1) + Dasatinib (Cycle 2, D1) | Vaccine + Dasatinib (Cycle 1, D1) | Total
Number analyzed (Participants) | 9 | 6 | 15
Age, Continuous [Mean (Full Range); unit: years] | 67.2 [44 to 75] | 64.7 [42 to 84] | 66.2 [42 to 84]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 3 | 7
  Male | 5 | 3 | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 9 | 6 | 15
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Stage of Disease [Count of Participants; unit: Participants] — NCI Cancer Staging:
  Stage 0: Abnormal cells are present but have not spread to nearby tissue. Also called carcinoma in situ, or CIS. CIS is not cancer, but it may become cancer.
  Stage I, Stage II, and Stage III: Cancer is present. The higher the number, the larger the cancer tumor and the more it has spread into nearby tissues.
  Stage IV: The cancer has spread to distant parts of the body.
  Participants
    Stage IIC | 0 | 1 | 1
    Stage IV | 8 | 5 | 13
    Not evaluable | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Immune Response Rate
Description: Immune Response is defined as improved peripheral blood CD8+ T cell responses against 3 or more peptide epitopes after active vaccination with Type I-polarized autologous dendritic cell (αDC1) vaccine incorporating 6 tumor blood vessel-associated antigen (TBVA)-derived peptides.
  The measure of Immune Response for this study is expressed as a proportion of responders: The number of HLA-A2+ melanoma patients with improved peripheral blood CD8+ T cell responses (responders) divided by the total number of evaluable patients.
Time Frame: Up to 13 months
Population: Patients that received at least one cycle of study treatment.
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Vaccine (Cycle 1, Day 1) + Dasatinib (Cycle 2, D1) | Vaccine + Dasatinib (Cycle 1, D1)
Number analyzed (Participants) | 7 | 6
proportion of participants | 0.29 [0.04 to 0.71] | 0.67 [0.22 to 0.96]

2. Secondary Outcome: Best Clinical Response
Description: The number of treated patients by best clinical response achieved (tumor measurements via radiologic evaluation) using RECIST 1.1. Complete Response (CR): Disappearance of all target lesions. Any pathological lymph nodes (target or non-target) with reduction in short axis to <10 mm. Partial Response (PR): ≥30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters. Stable Disease (SD): Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum diameters while on study. Progressive Disease (PD):≥20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). The sum must also demonstrate an absolute increase of ≥5 mm. The appearance ≥1 new lesion(s) is considered progression.
Time Frame: Up to 13 months
Population: Patients that received at least once cycle of study treatment who were evaluable for response using tumor measurements via radiologic evaluation.
Measure: Count of Participants; unit: Participants
Arm/Group | Vaccine (Cycle 1, Day 1) + Dasatinib (Cycle 2, D1) | Vaccine + Dasatinib (Cycle 1, D1)
Number analyzed (Participants) | 7 | 6
Participants
  Partial Response | 0 | 4
  Progressed Disease | 4 | 2
  Stable Disease | 3 | 0

3. Secondary Outcome: Objective Response Rate (ORR)
Description: The proportion of evaluable patients that achieved either partial or complete responses. Calculation: The number of patients who experienced a Partial Response (PR) + the number of patients who experienced a Complete Response (CR) / total number of response-evaluable patients.
  Per RECIST v1.1, Complete Response (CR): Disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm. Partial Response (PR): At least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters.
Time Frame: Up to 13 months
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Vaccine (Cycle 1, Day 1) + Dasatinib (Cycle 2, D1) | Vaccine + Dasatinib (Cycle 1, D1)
Number analyzed (Participants) | 7 | 6
proportion of participants | 0 [0 to 0.4096] | 0.6667 [0.2228 to 0.9567]

4. Secondary Outcome: Worst Grade of Any Toxicity
Description: Number of participants and severity grades for treatment-relatedness scores of possibly, probably, or definitely.
Time Frame: Up to 2 years
Population: Patients that received at least one dose of study treatment who experienced a treatment-related toxicity .
Measure: Count of Participants; unit: Participants
Arm/Group | Vaccine (Cycle 1, Day 1) + Dasatinib (Cycle 2, D1) | Vaccine + Dasatinib (Cycle 1, D1)
Number analyzed (Participants) | 9 | 6
Participants
  Grade 2 Toxicity | 1 | 2
  Grade 3 Toxicity | 6 | 3
  Grade 4 Toxicity | 0 | 1
  Grade 5 Toxicity | 1 | 0
  No >Grade 2 Toxicity | 1 | 0

5. Secondary Outcome: Progression-free Survival (PFS)
Description: The length of time after study treatment that a patient lives with disease but the disease does not progress. Patients were followed for 1 year after removal from study treatment or until death, whichever occurs first. Per RECIST 1.1, Progressive Disease is defined as a ≥ 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). The sum must also demonstrate an absolute increase of ≥5 mm. The appearance ≥1 new lesion(s) is considered progression.
Time Frame: Up to 15 months
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Vaccine (Cycle 1, Day 1) + Dasatinib (Cycle 2, D1) | Vaccine + Dasatinib (Cycle 1, D1)
Number analyzed (Participants) | 9 | 6
months | 1.967 [1.9 to NA] — Upper bound of the CI not reached | 7.867 [2.133 to NA] — Upper bound of the CI not reached

6. Secondary Outcome: Overall Survival (OS)
Description: The length of time from the start of study treatment, that patients remain alive.
Time Frame: Up to 30 months
Population: All patients enrolled in the study.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Vaccine (Cycle 1, Day 1) + Dasatinib (Cycle 2, D1) | Vaccine + Dasatinib (Cycle 1, D1)
Number analyzed (Participants) | 9 | 6
months | 3.667 [2.967 to NA] — Upper bound of CI not reached. | 17.83 [11.5 to NA] — Upper bound of CI not reached.

7. Secondary Outcome: T Cell-recruiting Chemokine CXCL10/IP-10
Description: Circulating serum concentration (levels) of T cell-recruiting chemokine CXCL10/IP-10 analyzed via ELISA assay. Higher levels of T cell-recruiting chemokine CXCL10/IP-1 correlate with patients exhibiting objective clinical response immunotherapy.
Time Frame: At baseline (prior to treatment)
Population: Patients that received Vaccine (Cycle 1, Day 1) + dasatinib (Cycle 2, D1) or Vaccine + dasatinib (both agents beginning Cycle 1, D1) for which there was an analyzable PBMC sample.
Measure: Mean (Full Range); unit: pg/mL
Arm/Group | Vaccine (Cycle 1, Day 1) + Dasatinib (Cycle 2, D1) | Vaccine + Dasatinib (Cycle 1, D1)
Number analyzed (Participants) | 7 | 6
pg/mL | 296.68 [120.04 to 931.2] | 268.06 [123.58 to 466.9]

8. Secondary Outcome: T Cell-recruiting Chemokine CXCL10/IP-10
Description: as for outcome 7
Time Frame: At between 5 and 7 weeks, post treatment
Population: as for outcome 7
Measure: Mean (Full Range); unit: pg/mL
Arm/Group | Vaccine (Cycle 1, Day 1) + Dasatinib (Cycle 2, D1) | Vaccine + Dasatinib (Cycle 1, D1)
Number analyzed (Participants) | 7 | 6
pg/mL | 501.43 [152.96 to 1889.6] | 194.96 [80.61 to 360.0]

9. Secondary Outcome: Treg CD4FoxP3 Suppressor Cells
Description: Percentage of Treg CD4FoxP3 suppressor cells in patients' peripheral blood. The accumulation of Treg CD4FoxP3 suppressor cell populations correlates with tumor progression (disease progression) and negative prognosis.
Time Frame: At baseline (prior to treatment)
Population: as for outcome 7
Measure: Mean (Full Range); unit: percentage of cells
Arm/Group | Vaccine (Cycle 1, Day 1) + Dasatinib (Cycle 2, D1) | Vaccine + Dasatinib (Cycle 1, D1)
Number analyzed (Participants) | 7 | 6
percentage of cells | 6.67 [3.72 to 9.05] | 8.04 [2.16 to 17]

10. Secondary Outcome: Treg CD4FoxP3 Suppressor Cells
Description: as for outcome 9
Time Frame: At between 4 and 6 weeks, post treatment
Population: as for outcome 7
Measure: Mean (Full Range); unit: percentage of cells
Arm/Group | Vaccine (Cycle 1, Day 1) + Dasatinib (Cycle 2, D1) | Vaccine + Dasatinib (Cycle 1, D1)
Number analyzed (Participants) | 7 | 6
percentage of cells | 8.06 [4.21 to 16.9] | 6.27 [0.417 to 14.2]

11. Secondary Outcome: Treg CD4FoxP3 Suppressor Cells
Description: as for outcome 9
Time Frame: At between 7 and 10 weeks, post treatment
Population: as for outcome 7
Measure: Mean (Full Range); unit: percentage of cells
Arm/Group | Vaccine (Cycle 1, Day 1) + Dasatinib (Cycle 2, D1) | Vaccine + Dasatinib (Cycle 1, D1)
Number analyzed (Participants) | 7 | 6
percentage of cells | 7.38 [3.78 to 14.1] | 6.6 [0.282 to 20.5]

12. Secondary Outcome: Monocytic Myeloid Derived Suppressor Cells (M-MDSC)
Description: Percentage of Monocytic Myeloid Derived Suppressor Cells (M-MDSC) present in patients' peripheral blood. The accumulation of M-MDSC populations correlates with tumor progression (disease progression) and negative prognosis.
Time Frame: At baseline (prior to treatment)
Population: as for outcome 7
Measure: Mean (Full Range); unit: percentage of cells
Arm/Group | Vaccine (Cycle 1, Day 1) + Dasatinib (Cycle 2, D1) | Vaccine + Dasatinib (Cycle 1, D1)
Number analyzed (Participants) | 7 | 6
percentage of cells | 6.23 [2.65 to 10.4] | 11.65 [0.707 to 23.4]

13. Secondary Outcome: Monocytic Myeloid Derived Suppressor Cells (M-MDSC)
Description: as for outcome 12
Time Frame: At between 4 and 6 weeks, post treatment
Population: as for outcome 7
Measure: Mean (Full Range); unit: percentage of cells
Arm/Group | Vaccine (Cycle 1, Day 1) + Dasatinib (Cycle 2, D1) | Vaccine + Dasatinib (Cycle 1, D1)
Number analyzed (Participants) | 7 | 6
percentage of cells | 8.7 [3.29 to 12.6] | 8.78 [2.59 to 20.6]

14. Secondary Outcome: Monocytic Myeloid Derived Suppressor Cells (M-MDSC)
Description: as for outcome 12
Time Frame: At between 7 and 10 weeks, post treatment
Population: as for outcome 7
Measure: Mean (Full Range); unit: percentage of cells
Arm/Group | Vaccine (Cycle 1, Day 1) + Dasatinib (Cycle 2, D1) | Vaccine + Dasatinib (Cycle 1, D1)
Number analyzed (Participants) | 7 | 6
percentage of cells | 9.32 [0.131 to 24.6] | 8.32 [0.433 to 17.2]

15. Secondary Outcome: Polymorphonucler Myeloid-derived Suppressor Cells (PMN-MDSC)
Description: Percentage of Polymorphonucler myeloid-derived suppressor cells (PMN-MDSC) present in patients' peripheral blood. The accumulation/increase of M-MDSC populations correlates with tumor progression (disease progression) and negative prognosis.
Time Frame: At baseline (prior to treatment)
Population: as for outcome 7
Measure: Mean (Full Range); unit: percentage of cells
Arm/Group | Vaccine (Cycle 1, Day 1) + Dasatinib (Cycle 2, D1) | Vaccine + Dasatinib (Cycle 1, D1)
Number analyzed (Participants) | 7 | 6
percentage of cells | 12.36 [5.02 to 20.1] | 11.59 [1.24 to 23]

16. Secondary Outcome: Polymorphonucler Myeloid-derived Suppressor Cells (PMN-MDSC)
Description: as for outcome 15
Time Frame: At between 4 and 6 weeks, post treatment
Population: as for outcome 7
Measure: Mean (Full Range); unit: percentage of cells
Arm/Group | Vaccine (Cycle 1, Day 1) + Dasatinib (Cycle 2, D1) | Vaccine + Dasatinib (Cycle 1, D1)
Number analyzed (Participants) | 7 | 6
percentage of cells | 10.14 [3.39 to 14.4] | 14.61 [0.865 to 49.7]

17. Secondary Outcome: Polymorphonucler Myeloid-derived Suppressor Cells (PMN-MDSC)
Description: as for outcome 15
Time Frame: At between 7 and 10 weeks, post treatment
Population: as for outcome 7
Measure: Mean (Full Range); unit: percentage of cells
Arm/Group | Vaccine (Cycle 1, Day 1) + Dasatinib (Cycle 2, D1) | Vaccine + Dasatinib (Cycle 1, D1)
Number analyzed (Participants) | 7 | 6
percentage of cells | 9.41 [2.46 to 23.5] | 12.45 [1.08 to 26.7]

18. Secondary Outcome: EphA2 Protein Expression in Tumor Biopsies
Description: Level of EphA2 protein expression in tumor tissue biopsies.
Time Frame: Up to 6 months
Population: Results not achievable due to insufficient patient biopsy material for the assays required for this endpoint.
Arm/Group | Vaccine (Cycle 1, Day 1) + Dasatinib (Cycle 2, D1) | Vaccine + Dasatinib (Cycle 1, D1)
Number analyzed (Participants) | 0 | 0

19. Secondary Outcome: Suppressor Cell Populations and Blood Vessels in Melanoma Tumor Biopsies
Description: Percentage of suppressor cell populations and blood vessels in melanoma tumor biopsies.
Time Frame: Up to 6 months
Population: Results not achievable due to insufficient patient biopsy material for the assays required for this endpoint.
Arm/Group | Vaccine (Cycle 1, Day 1) + Dasatinib (Cycle 2, D1) | Vaccine + Dasatinib (Cycle 1, D1)
Number analyzed (Participants) | 0 | 0

20. Secondary Outcome: CD8+ T Cells Infiltration
Description: Percentage of CD8+ T cells infiltrating into melanoma lesions (tumor tissues).
Time Frame: Up to 6 months
Population: Results not achievable due to insufficient patient biopsy material for the assays required for this endpoint.
Arm/Group | Vaccine (Cycle 1, Day 1) + Dasatinib (Cycle 2, D1) | Vaccine + Dasatinib (Cycle 1, D1)
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Up to 3 years
Description: This study will use the CTCAE (Common Terminology Criteria for Adverse Events) version 4.0. for toxicity and serious adverse event reporting. Adverse Events will be evaluated and data collected from Week 1 through Week 8 during treatment, up to and during the off study treatment visit.
Arm/Group | Vaccine (Cycle 1, Day 1) + Dasatinib (Cycle 2, D1) | Vaccine + Dasatinib (Cycle 1, D1)
All-Cause Mortality (participants affected / at risk) | 8/9 | 5/6
Serious Adverse Events (participants affected / at risk) | 7/9 | 4/6
Other Adverse Events (participants affected / at risk) | 8/9 | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Vaccine (Cycle 1, Day 1) + Dasatinib (Cycle 2, D1) (N=9) | Vaccine + Dasatinib (Cycle 1, D1) (N=6)
Anemia (Blood and lymphatic system disorders) | 1 | 2
Cardiac disorders - Other, specify (Cardiac disorders) | 0 | 1
Adrenal insufficiency (Endocrine disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 2 | 0
Constipation (Gastrointestinal disorders) | 1 | 0
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0
Fatigue (General disorders) | 1 | 0
Gait disturbance (General disorders) | 0 | 1
Non-cardiac chest pain (General disorders) | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 1
Investigations - Other, specify (Investigations) | 1 | 0
Lymphocyte count decreased (Investigations) | 2 | 0
Urine output decreased (Investigations) | 0 | 1
Anorexia (Metabolism and nutrition disorders) | 0 | 1
Hyperuricemia (Metabolism and nutrition disorders) | 1 | 0
Hypophosphatemia (Metabolism and nutrition disorders) | 0 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Encephalopathy (Nervous system disorders) | 0 | 1
Confusion (Psychiatric disorders) | 1 | 1
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 0
Hypotension (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Vaccine (Cycle 1, Day 1) + Dasatinib (Cycle 2, D1) (N=9) | Vaccine + Dasatinib (Cycle 1, D1) (N=6)
Anemia (Blood and lymphatic system disorders) | 5 | 3
Leukocytosis (Blood and lymphatic system disorders) | 0 | 1
Palpitations (Cardiac disorders) | 1 | 0
Sinus tachycardia (Cardiac disorders) | 1 | 1
Ear pain (Ear and labyrinth disorders) | 0 | 1
Endocrine disorders - Other, specify (Endocrine disorders) | 0 | 1
Hypoparathyroidism (Endocrine disorders) | 0 | 1
Hypothyroidism (Endocrine disorders) | 0 | 2
Eyelid function disorder (Eye disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 2
Constipation (Gastrointestinal disorders) | 1 | 0
Diarrhea (Gastrointestinal disorders) | 2 | 3
Dry mouth (Gastrointestinal disorders) | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 0 | 2
Dysphagia (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 1 | 5
Vomiting (Gastrointestinal disorders) | 0 | 4
Chills (General disorders) | 2 | 1
Edema limbs (General disorders) | 0 | 1
Fatigue (General disorders) | 5 | 5
Fever (General disorders) | 2 | 2
Malaise (General disorders) | 1 | 0
General disorders and administration site conditions - Other, specify (General disorders) | 0 | 3
Non-cardiac chest pain (General disorders) | 0 | 1
Pain (General disorders) | 3 | 2
Eye infection (Infections and infestations) | 0 | 1
Infections and infestations - Other, specify (Infections and infestations) | 0 | 2
Lung infection (Infections and infestations) | 1 | 0
Lymph gland infection (Infections and infestations) | 0 | 1
Phlebitis infective (Infections and infestations) | 0 | 1
Skin infection (Infections and infestations) | 1 | 0
Upper respiratory infection (Infections and infestations) | 1 | 1
Urinary tract infection (Infections and infestations) | 1 | 0
Bruising (Injury, poisoning and procedural complications) | 0 | 1
Activated partial thromboplastin time prolonged (Investigations) | 0 | 1
Alkaline phosphatase increased (Investigations) | 3 | 1
Aspartate aminotransferase increased (Investigations) | 2 | 3
Cardiac troponin I increased (Investigations) | 0 | 1
Creatinine increased (Investigations) | 0 | 2
Investigations - Other, specify (Investigations) | 0 | 3
Investigations - Other, specify (Investigations) | 3 | 0
Lymphocyte count decreased (Investigations) | 2 | 3
Neutrophil count decreased (Investigations) | 2 | 4
Platelet count decreased (Investigations) | 2 | 3
Weight loss (Investigations) | 1 | 1
White blood cell decreased (Investigations) | 1 | 2
Anorexia (Metabolism and nutrition disorders) | 3 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 1
Hyperglycemia (Metabolism and nutrition disorders) | 0 | 2
Hypermagnesemia (Metabolism and nutrition disorders) | 0 | 1
Hypoalbuminemia (Metabolism and nutrition disorders) | 4 | 4
Hypocalcemia (Metabolism and nutrition disorders) | 2 | 2
Hypoglycemia (Metabolism and nutrition disorders) | 0 | 2
Hypokalemia (Metabolism and nutrition disorders) | 1 | 2
Hypomagnesemia (Metabolism and nutrition disorders) | 1 | 0
Hyponatremia (Metabolism and nutrition disorders) | 5 | 5
Hypophosphatemia (Metabolism and nutrition disorders) | 2 | 2
Metabolism and nutrition disorders - Other, specify (Metabolism and nutrition disorders) | 2 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 1 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 3
Dizziness (Nervous system disorders) | 3 | 2
Dysarthria (Nervous system disorders) | 0 | 1
Headache (Nervous system disorders) | 1 | 4
Hallucinations (Psychiatric disorders) | 1 | 1
Insomnia (Psychiatric disorders) | 0 | 3
Psychiatric disorders - Other, specify (Psychiatric disorders) | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 1 | 0
Bladder spasm (Renal and urinary disorders) | 1 | 1
Uterine hemorrhage (Reproductive system and breast disorders) | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 2
Erythema multiforme (Skin and subcutaneous tissue disorders) | 1 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 2
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 3
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 1 | 2
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 1
Hot flashes (Vascular disorders) | 1 | 0
Hypertension (Vascular disorders) | 0 | 1
Lymphedema (Vascular disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-07-14): https://cdn.clinicaltrials.gov/large-docs/12/NCT01876212/Prot_SAP_000.pdf